CLINICAL TRIAL: NCT00668044
Title: A Population Pharmacokinetics Study of Plasma Levels of Ciprofloxacin Following a Regimen of Repeated Dose I.V. Administration (400 mg TID) on Burn Patients
Brief Title: Ciprofloxacin on Burned Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer HealthCare AG
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10627; COB
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-10

CONDITIONS: Burns; Bacterial Infections
Keywords: Ciprofloxacin regimen in compromised patients; Ciprofloxacin; Burned patients
MeSH Terms: conditions — Burns; Bacterial Infections | interventions — Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Ciprofloxacin (BAYO9867)
- Arm 2 (Experimental)
  Interventions: Drug: Ciprofloxacin (BAYO9867)

INTERVENTIONS:
Drug: Ciprofloxacin (BAYO9867) — 400 mg iv BID
  Arms: Arm 1
Drug: Ciprofloxacin (BAYO9867) — 400 mg iv TID
  Arms: Arm 2

SUMMARY:
This was a non randomised, multi center, italian study performed in burn patients receiving an antibiotic (ciprofloxacin) in order to treat an active infection. The aim of the study was to validate a pharmacokinetics model useful to verify if a standard dose regimen of ciprofloxacin, given to patients with a compromised metabolism, is a correct dose or instead is over or under dosed.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe burnt patients defined as burning of 20 to 60% of total body surface according to rule of nine, II deep degree and III degree according to Full-Thickness Burn model,
* Hospitalization for burning injury since at least 72h during hyper metabolic phase
* Active infections microbiological confirmed
* Signed informed consent

Exclusion Criteria:

* Pregnant or lactating female patients
* Previous history of tendinopathy
* Knowing syndrome of QTc prolongation
* Impairment renal function
* Hepatic insufficiency
* Convulsion
* Limited life expectancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2002-11; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Achievement of a population mean plasma level/time profile for the 400mg i.v. ciprofloxacin aimed to validate a pk model | >72 h post injury, 48h and 120 h after treatment

SECONDARY OUTCOMES:
Evaluation of AreaUnderCurve/Minimal Inhibiting Concentration Ratio | >72 h post injury, 48h and 120 h after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (6):
- Italy (6):
  - Cesena, Forlì
  - Catania
  - Genova
  - Padua
  - Palermo
  - Roma